CLINICAL TRIAL: NCT04096404
Title: A Longitudinal Study to Determine the Effect of Gene-based Personalised Diet and Physical Activity Advice on Adiposity Indices in University Students
Brief Title: Gene-based Personalised Diet and Physical Activity Advice on Adiposity Indices Personalised Diet and Physical Activity Advice on Adiposity Indices in University Students
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: St Mary's University College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SMEC_2018-19_052
Record Dates: First submitted 2019-08-16; First posted 2019-09-19 (Actual); Last update posted 2019-09-19 (Actual); Status verified 2019-09

CONDITIONS: Adiposity; Behavior, Health
MeSH Terms: conditions — Obesity; Health Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): no advice
- Non genetic personalised advice (Active Comparator): dietary and physical activity advice based on reported dietary intake and physical activity
  Interventions: Behavioral: Non genetic personalised advice
- Genotype- based personalised advice (Experimental): dietary and physical activity advice based on genotype, reported dietary intake and physical activity
  Interventions: Genetic: Genotype- based personalised advice; Behavioral: Non genetic personalised advice

INTERVENTIONS:
Genetic: Genotype- based personalised advice — Following allocation to groups participants will receive appropriate dietary and physical activity advice based on their genotype via email
  Arms: Genotype- based personalised advice
Behavioral: Non genetic personalised advice — Following allocation to groups participants will receive appropriate dietary and physical activity advice based on their reported intake, BMI and activity via email
  Arms: Genotype- based personalised advice; Non genetic personalised advice

SUMMARY:
A longitudinal study to determine the effect of gene-based personalised diet and physical activity advice on adiposity indices in university students.

DETAILED DESCRIPTION:
The study uses a randomised controlled design; data for all variables (participant characteristics, height, weight, body mass index (BMI), waist circumference (WC), body fat percentage (BF%), healthy eating motivation, dietary intake and physical activity) will be collected initially from participants at St Mary's University during September and October 2019. Participants will be genotyped, stratified randomisation (based on genotype and BMI) will be used to allocate participants to three different groups (1. Control: no advice, 2. Non genetic personalised advice: dietary and physical activity advice based on reported dietary intake and physical activity 3. Genotype- based personalised advice: dietary and physical activity advice based on genotype, reported dietary intake and physical activity. Following allocation to groups participants in groups 2 and 3 will receive appropriate dietary and physical activity advice via email (appendix a) and all participants will complete the healthy eating motivation questionnaire for a second time. In April/May 2020 follow up variables (smoking status, weight, BMI, WC, BF%, healthy eating motivation, dietary intake and physical activity) will be measured again. These follow up variables will be measured every September and April/May until September 2022. After each follow up participants in groups 2 and 3 will be resent their dietary and physical activity advice and updated information based on their reported dietary intake and physical activity.

ELIGIBILITY:
Inclusion Criteria:

• Age 18-25 years

Exclusion Criteria:

* Pregnancy and lactation
* Chronic disease
* A history of disordered eating and following a restricted diet.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 400 (Estimated)
Dates: Start 2019-09 (Estimated); Primary Completion 2022-09 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Body weight in kg | 3 years
  Weight will be measured to the nearest 0.1 kg
Body fat percentage | 3 years
  Body fat percentage will be measured to the nearest 0.1%
Body mass index in Kg/m2 | 3 years
  calculated from measured height and weight

SECONDARY OUTCOMES:
Dietary intake | 3 years
  using a four day food diary collected using a food diary and nutritional analysis app (Libro, 2018)
Physical activity | 3 years
  using the Epic Physical Activity Questionnaire (EPAQ2) (Wareham et al., 2002)
Participants motivation to eat healthily | 3 years
  measured using the Healthy Eating Motivation Score (Naughton et al., 2015)

IPD SHARING:
Plan to Share IPD: No